CLINICAL TRIAL: NCT00882050
Title: Intravenous Exenatide (Byetta) for the Treatment of Perioperative Hyperglycemia: Rollover Phase I/II Trial
Brief Title: Intravenous Exenatide (Byetta) During Surgery
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Thomas Jefferson University (Other)
Collaborators: Amylin Pharmaceuticals, LLC. (Industry); Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 808104
Record Dates: First submitted 2009-04-15; First posted 2009-04-16 (Estimated); Results first posted 2022-01-21 (Actual); Last update posted 2022-01-21 (Actual); Status verified 2021-12

CONDITIONS: Euglycemia; Hypoglycemia; Hyperglycemia
MeSH Terms: conditions — Hypoglycemia; Hyperglycemia | interventions — Exenatide; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Exentatide 0.27 ng/kg/min (Experimental): Exenatide to be infused by intravenous method at 0.27 ng/kg/min (0.066 pmol/kg/min) over 3-6 hours.
  * Induction of anesthesia will be equal to Intubation time. Infusion will begin at this time point (+ or - 3 minutes).
  * Blood samples will be obtained prior to intubation and then 10 and 30 minutes after drug initiation and every 30 minutes (+ or - 2 minutes) thereafter until the infusion is stopped. The drug infusion will be stopped at extubation. Blood will then be sampled every 30 minutes (+ or - 2 minutes) post extubation for 2 hours, and once 24 hours after extubation.
  * Blood plasma levels will be collected (8-10 mls) for analysis of GLP-1, Glucose, Potassium, Insulin, Glucagon, Epinephrine, Norepinephrine, Cortisol, and free fatty acids (FFA).
  Interventions: Drug: Exenatide 0.27 ng/kg/min
- Exentatide 0.41 ng/kg/min (Experimental): Experimental: IV Exenatide to be infused by intravenous method at 0.41 ng/kg/min (0.099 pmol/kg/min) over 3 to 6 hours.
  * Induction of anesthesia will be equal to Intubation time. Infusion will begin at this time point (+ or - 3 minutes).
  * Blood samples will be obtained prior to intubation and then 10 and 30 minutes after drug initiation and every 30 minutes (+ or - 2 minutes) thereafter until the infusion is stopped. The drug infusion will be stopped at extubation. Blood will then be sampled every 30 minutes (+ or - 2 minutes) post extubation for 2 hours, and once 24 hours after extubation.
  * Blood plasma levels will be collected (8-10 mls) for analysis of GLP-1, Glucose, Potassium, Insulin,Glucagon, Epinephrine, Norepinephrine, Cortisol, and free fatty acids (FFA).
  Interventions: Drug: Exenatide 0.41 ng/kg/min
- Placebo IV NSS (Placebo Comparator): Placebo of IV normal saline solution as comparator.
  * Induction of anesthesia will be equal to Intubation time. Infusion will begin at this time point (+ or - 3 minutes).
  * Blood samples will be obtained prior to intubation and then 10 and 30 minutes after drug initiation and every 30 minutes (+ or - 2 minutes) thereafter until the infusion is stopped. The drug infusion will be stopped at extubation. Blood will then be sampled every 30 minutes (+ or - 2 minutes) post extubation for 2 hours, and once 24 hours after extubation.
  * Blood plasma levels will be collected (8-10 mls) for analysis of GLP-1, Glucose, Potassium, Insulin, Glucagon, Epinephrine, Norepinephrine, Cortisol, and free fatty acids (FFA).
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Exenatide 0.27 ng/kg/min — Exenatide to be infused intravenously at 0.27 ng/kg/min (0.066 pmol/kg/min) for a duration of 3 to 6 hours.
  * Induction of anesthesia will be equal to Intubation time. Infusion will begin at this time point (+ or - 3 minutes).
  * Blood samples will be obtained prior to intubation and then 10 and 30 minutes after drug initiation and every 30 minutes (+ or - 2 minutes) thereafter until the infusion is stopped. The drug infusion will be stopped at extubation. Blood will then be sampled every 30 minutes (+ or - 2 minutes) post extubation for 2 hours, and once 24 hours after extubation.
  * Blood plasma levels will be collected (8-10 mls) for analysis of GLP-1, Glucose, Potassium, Insulin, Glucagon, Epinephrine, Norepinephrine, Cortisol, and free fatty acids (FFA).
  Other Names: Byetta
  Arms: Exentatide 0.27 ng/kg/min
Drug: Exenatide 0.41 ng/kg/min — Exenatide to be infused intravenously 0.41 ng/kg/min (0.099 pmol/kg/min) for a duration of 3 to 6 hours Induction of anesthesia will be equal to Intubation time. Infusion will begin at this time point (+ or - 3 minutes).
  * Blood samples will be obtained prior to intubation and then 10 and 30 minutes after drug initiation and every 30 minutes (+ or - 2 minutes) thereafter until the infusion is stopped. The drug infusion will be stopped at extubation. Blood will then be sampled every 30 minutes (+ or - 2 minutes) post extubation for 2 hours, and once 24 hours after extubation.
  * Blood plasma levels will be collected (8-10 mls) for analysis of GLP-1, Glucose, Potassium, Insulin, Glucagon, Epinephrine, Norepinephrine, Cortisol, and free fatty acids (FFA).
  Other Names: Byetta
  Arms: Exentatide 0.41 ng/kg/min
Drug: Placebo — Intravenous Placebo of NSS infused at same rate as drug comparator. Induction of anesthesia will be equal to Intubation time. Infusion will begin at this time point (+ or - 3 minutes).
  * Blood samples will be obtained prior to intubation and then 10 and 30 minutes after drug initiation and every 30 minutes (+ or - 2 minutes) thereafter until the infusion is stopped. The drug infusion will be stopped at extubation. Blood will then be sampled every 30 minutes (+ or - 2 minutes) post extubation for 2 hours, and once 24 hours after extubation.
  * Blood plasma levels will be collected (8-10 mls) for analysis of GLP-1, Glucose, Potassium, Insulin, Glucagon, Epinephrine, Norepinephrine, Cortisol, and free fatty acids (FFA).
  Other Names: Normal Saline Solution
  Arms: Placebo IV NSS

SUMMARY:
The purpose of this project is to study if intravenous Exenatide is effective at maintaining normal blood glucose levels and preventing low blood glucose levels during surgery.

DETAILED DESCRIPTION:
This is a single-center, block randomized, double-blind, placebo-controlled, dose-ranging study. Subjects will be randomized in equal proportions to one of three treatment arms: placebo of normal saline solution, 0.27 ng/kg/min (0.066 pmol/kg/min) IV Exenatide, and 0.41 ng/kg/min (0.099 pmol/kg/min) IV Exenatide. We will use a block number of 30 (please see power analysis) so that balance between each of the three groups will be maintained over the enrollment period. We will stratify the randomization scheme to ensure balance of diabetics and non-diabetics within the groups.

ELIGIBILITY:
Inclusion Criteria:

* Age (>18 years)
* Weight of > 50 kg and < 150 kg
* Ability to provide informed consent
* Elective surgery including:
* Cardiac surgery to include elective CABG with or without single or multivalve repair or replacement and/or single or multivalve repair/replacement requiring CPB and sternotomy (to include subjects who are undergoing first time or redo cardiac surgery)
* Abdominal aortic aneurysm repair
* Carotid endarterectomy
* Esophagectomy
* Cystectomy
* Nephrectomy
* If female, subject must be non-lactating, and, if of childbearing potential, must have a negative urine pregnancy test within 24 hours prior to receiving study drug

Exclusion Criteria:

* Age (<18 years)
* Inability to provide informed consent
* History or risk of pancreatitis (e.g. ethanol abuse, gall stones)
* Receipt of an investigational drug or device with 30 days prior to surgery
* Use of any concomitant medication listed above on the day of surgery
* Known allergy to Exenatide, fentanyl, midazolam, isoflurane, propofol, heparin or neuromuscular blockers
* Known substance abuse
* Surgical procedure other than:

Cardiac surgery to include elective CABG with or without single or multivalve repair or replacement and/or single or multivalve repair/ replacement requiring CPB and sternotomy (to include subjects who are undergoing first time or redo cardiac surgery)

* Abdominal aortic aneurysm repair
* Carotid endarterectomy
* Esophagectomy
* Cystectomy
* Nephrectomy

  * Insulin dependent diabetes mellitis
  * Anticipated administration of intraoperative steroids
  * Major end organ dysfunction, defined as:
* Current intravenous inotropic agents
* Preoperative use of intra-aortic balloon pump (IABP), left ventricular assist device (LVAD), or extracorporeal membrane oxygenation (ECMO)
* Renal
* Preoperative serum Creatinine > 2.0 mg/dL
* Hepatic
* History of abnormal hepatic function in the past
* Hematologic
* Preoperative hematocrit (HCT) < 30%
* Platelet count < 100,000/mm3
* History of bleeding or clotting disorder

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 104 (Actual)
Dates: Start 2009-03; Primary Completion 2016-04 (Actual); Study Completion 2016-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Benjamin A. Kohl, MD, Study Director — University of Pennsylvania
Locations (1):
- University of Pennsylvania, Philadelphia, Pennsylvania, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Screening started in the appropriate surgical clinic on 3/29/2009 and continued until 5/14/2012 when Dr. Ben Kohl was recruited away from Penn. Recruitment resumed with Dr. Prakash Patel on 9/22/14 and ended 3/20/2015. During active enrollment 104 subjects were enrolled and an additional 96 potential subjects failed screening or declined.
Groups:
- Exentatide 0.27 ng/kg/Min: Exenatide IV 0.27 ng/kg/min (0.066 pmol/kg/min) over 3-6 hours. Induction of anesthesia will be equal to intubation time and drug will start (+ or-3 min).
  * Blood will be collected prior to intubation and then 10 and 30 min after drug initiation and every 30 min (+or-2 min) until the IV is stopped and/or at extubation. Sample collection every 30 min post extubation for 2 hours, and once at 24 hours after extubation.
  * Analysis of GLP-1, Glucose, Potassium, Insulin, Glucagon, Epinephrine, Norepinephrine, Cortisol, and free fatty acids (FFA) will be conducted.
Period: Overall Study
Arm/Group | Exentatide 0.27 ng/kg/Min | Exentatide 0.41 ng/kg/Min | Placebo IV NSS
Started | 32 | 33 | 39
Completed | 31 | 33 | 39
Not Completed | 1 | 0 | 0
Not completed — Physician Decision | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Exentatide 0.27 ng/kg/Min: Demographics Exen 0.27 ng/kg/min
  Sex: Female 9 Male 23 Age , mean (SD) 64.1 (13.41) Race: African American: 2 Caucasian: 30 Ethnicity: Non-Hispanic 32
- Exentatide 0.41 ng/kg/Min: Table 1: Demographics Exen 0.41 ng/kg/min
  Sex: Female 13 Male 20 Age , mean (SD) 67.4 (11.98) Race: African American: 2 Caucasian: 31 Ethnicity: Non-Hispanic 33
- Placebo of IV NSS: Table 1: Demographics placebo Sex: Female 11 Male 28 Age, mean (SD) 66.2 (13.56) Race: African American: 5 Caucasian: 34 Ethnicity: Non-Hispanic 39
- Total: Total of all reporting groups
Arm/Group | Exentatide 0.27 ng/kg/Min | Exentatide 0.41 ng/kg/Min | Placebo of IV NSS | Total
Number analyzed (Participants) | 32 | 33 | 39 | 104
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 14 | 12 | 18 | 44
  >=65 years | 18 | 21 | 21 | 60
Age, Continuous [Mean (Full Range); unit: years] | 64.1 [26 to 84] | 67.4 [30 to 83] | 66.2 [39 to 86] | 65.9 [26 to 86]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 13 | 11 | 33
  Male | 23 | 20 | 28 | 71
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 2 | 2 | 5 | 9
  White | 30 | 31 | 34 | 95
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 32 | 33 | 39 | 104

OUTCOME MEASURES:

1. Primary Outcome: The Primary Objective is to Determine the Ability of Intravenous Exenatide to: Maintain Intraoperative Euglycemia in Subjects With Initial Blood Glucose < 126 mg/dL in Surgical Subjects as Compared to Placebo,
Description: Logistic regression analysis will be utizlized to determine maintenance of euglycemia (yes v no) for our primary analysis. A standard area under the curve (AUC) analysis will be performed for each time point to map out drug deposition. Assuming a standard 2 compartment model, 10 subjects per group is sufficient to accurately predict mean AUC. Our primary analysis should provide ample statistical power.
Time Frame: Baseline and 90 minutes after starting infusion;
Population: 104 subjects were enrolled. 39 subjects randomized to placebo, 32 in 0.27 ng/kg/min, and 33 to 41 ng/kg/minute. One subject was removed from the study at the request of the surgeon. No intraoperative blinded infusions (study drug) were discontinued in any other case.
Measure: Mean (Standard Deviation); unit: mlg/dL
Groups:
- Exentatide 0.27 ng/kg/Min: Experimental: IV Exenatide to be infused by intravenous method at 0.27 ng/kg/min (0.099 pmol/kg/min) over 3 to 6 hours. Minimum time of infusion 90 minutes.
- Exenatide 0.41ng/kg/Min: Experimental: IV Exenatide to be infused by intravenous method at 0.41 ng/kg/min (0.099 pmol/kg/min) over 3 to 6 hours. Minimum time of infusion 90 minutes.
- Placebo IV NSS: Placebo: IV NSS to be infused by intravenous method at rate for experimental drug over 3 to 6 hours. Minimum 90 minutes.
Arm/Group | Exentatide 0.27 ng/kg/Min | Exenatide 0.41ng/kg/Min | Placebo IV NSS
Number analyzed (Participants) | 32 | 33 | 39
mlg/dL
  Pre glucose levels | 112.3 (24.1) | 108.1 (27.8) | 110.4 (17.3)
  at 90 minutes post infusion glucose levels | 120.3 (36.3) | 125.0 (22.9) | 120.8 (29.7)
Statistical Analysis 1: Comparison: Exentatide 0.27 ng/kg/Min vs Exenatide 0.41ng/kg/Min vs Placebo IV NSS; logistic regression; Test type: Other; p = 0.05, Regression, Logistic; Because we tested interventions against the placebo arm, we increased our subjects to overcome loss of power. 23 per group will provide 80% power assuming a reduced alpha of 0.01 to accommodate the multiple testing issues
Statistical Analysis 2: Comparison: Exentatide 0.27 ng/kg/Min vs Exenatide 0.41ng/kg/Min vs Placebo IV NSS; Primary t tests of glucose between the 3 groups at 90 minutes post. Secondary MANOVA to determine the effect over time. Change in mean glucose of 20 mg/dl between all groups detectable by 18 subjects per group assuming a SD of 20mg/dl., an 82% power with an alpha of 0.05. Because we tested interventions against the placebo arm, we increased our subjects to overcome loss of power. 23 per group will provide 80% power assuming a reduced alpha of 0.01 to accommodate the multiple testing issues; Test type: Superiority — Demographic data analyzed with nominal data tested by chi-square, ordinal data by Mann-Whitney, and normal data by t-test. Further, a linear regression analysis to determine the effect of intervention dose on glucose level and typical confounders such as age, weight, and type of surgery was completed. Adverse and SAEs were analyzed by chi-square for occurrence; p = 0.05, Regression, Logistic — Due to have 3 trial groups our p value was adjusted for multiple comparisons as a a priori threshold (if a single comparison) was 0.05; The regression (see above) is a secondary analysis. Groups had been stratified on diabetic (y/n) to balance this potential confounder

ADVERSE EVENTS:
Time Frame: AEs were collected on each subject from time of signed consent until 24 hours post surgery. This time frame was approximately one month.
Description: Any untoward or unfavorable medical occurrence in a participant, including any abnormal sign (for example, abnormal physical exam or laboratory finding), symptom, or disease, temporally associated with the participant's participation in the research, whether or not considered related to the participant's participation in the research.
Groups:
- Exentatide 0.27 ng/kg/Min: Exenatide to be infused by intravenous method at 0.27 ng/kg/min (0.066 pmol/kg/min) over 3-6 hours. Minimum 90 minutes post infusion.
- Exenatide 0.41ng/kg/Min: Exenatide to be infused by intravenous method at 0.41 ng/kg/min (0.066 pmol/kg/min) over 3-6 hours. Minimum 90 minutes post infusion.
- Placebo IV NSS: Placebo IV NSS to be at the rate of the experimental groups over 3-6 hours. Minimum 90 minutes post infusion.
Arm/Group | Exentatide 0.27 ng/kg/Min | Exenatide 0.41ng/kg/Min | Placebo IV NSS
All-Cause Mortality (participants affected / at risk) | 0/32 | 0/33 | 0/39
Serious Adverse Events (participants affected / at risk) | 0/32 | 0/33 | 0/39
Other Adverse Events (participants affected / at risk) | 2/32 | 0/33 | 0/39
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Exentatide 0.27 ng/kg/Min (N=32) | Exenatide 0.41ng/kg/Min (N=33) | Placebo IV NSS (N=39)
Ischemia (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) — Study drug had infused about 1 hour when surgery was stopped due to concern of ischemia on telemetry (prior history). Subject was ruled out for myocardial infarction (3 sets cardiac enzymes negative). Released next day. Not related to study drug.
Left sided weakness (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) — Left sided weakness 30 hrs post op (AVR). Had CT scan & neurology consult. Probable subacute infarct in right frontal lobe. No significant mass effect, no hemorrhage. Subject monitored, recovered fully prior to discharge. Not related to study drug.

LIMITATIONS AND CAVEATS:
Change in PI during the trial led to intermittent study activitity and a delay in enrollment which prolonged the study and final data entry.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No